CLINICAL TRIAL: NCT00000486
Title: Unstable Angina Pectoris Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2000-01

CONDITIONS: Angina, Unstable; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia
MeSH Terms: conditions — Angina, Unstable; Cardiovascular Diseases; Coronary Disease; Heart Diseases; Myocardial Ischemia | interventions — Coronary Artery Bypass

INTERVENTIONS:
Procedure: coronary artery bypass

SUMMARY:
To compare the efficacy of medical or surgical (coronary artery bypass graft) therapy with regard to survival and quality of life in patients with unstable angina and requisite coronary anatomy as defined by angiography.

DETAILED DESCRIPTION:
BACKGROUND:

Angina pectoris is a symptomatic condition of attacks of chest pain, often debilitating. It is caused by a decreased supply of blood to the heart, such as that which might occur in coronary artery disease. The usual treatment of angina pectoris is designed to relieve the symptoms. It includes avoidance of activities that produce the discomfort and the use of nitroglycerin and beta blocking drugs. Soon after the introduction of coronary bypass surgery, many doctors enthusiastically adopted this approach in treating patients with unstable angina.

In 1972, emphasizing that there was no definitive evidence showing the superiority of intensive medical management or coronary bypass surgery in determining mortality and morbidity in patients hospitalized with unstable angina, some of the participating groups in the NHLBI Myocardial Infarction Research Units developed a cooperative clinical trial to compare these medical and surgical approaches to therapy.

From 1972 through 1976, 288 patients were entered into this randomized clinical trial. One hundred forty-seven patients received intensive pharmacological medical therapy, and 141 comparable patients underwent coronary artery bypass surgery. Careful follow-up studies were performed on patients in both groups, in-hospital and during the post-hospital phase. These studies included, apart from routine physical examinations, resting electrocardiograms, chest x-ray films, and grade exercise tolerance tests at six months and twelve months.

DESIGN NARRATIVE:

Randomized, non-blind, sequential design with a control group and an experimental group. The patients in the experimental group were treated with coronary bypass surgery. Patients in the control group received intensive medical management. Endpoints were mortality and morbidity measures, such as incidence of myocardial infarction and persistence of angina.

ELIGIBILITY:
Men and women, ages 21 to 65. Angina pectoris (class III or class IV) at rest or with minimal exercise.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1972-01; Study Completion 1980-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Becker — Johns Hopkins University; Adolph Hutter — Massachusetts General Hospital; Leon Resnekov — University of Chicago; Richard Russell — University of Alabama at Birmingham; John Schroeder — Stanford University; Andrew Wallace — Duke University

REFERENCES:
- [Background] Unstable angina pectoris: national cooperative study group to compare medical and surgical therapy. I. Report of protocol and patient population. Am J Cardiol. 1976 May;37(6):896-902. doi: 10.1016/0002-9149(76)90116-8. PMID 1266755
- [Background] Unstable angina pectoris: national cooperative study group to compare surgical and medical therapy. III. Results in patients with S-T segment elevation during pain. Am J Cardiol. 1980 Apr;45(4):819-24. doi: 10.1016/0002-9149(80)90127-7. No abstract available. PMID 6965816
- [Background] Russell RO Jr, Wayne JB, Kronefeld J, Charles ED, Oberman A, Kouchoukos NT, White C, Rogers W, Mantle JA, Rackley CE. Surgical versus medical therapy for treatment of unstable angina: changes in work status and family income. Am J Cardiol. 1980 Jan;45(1):134-40. doi: 10.1016/0002-9149(80)90231-3. No abstract available. PMID 6965333